CLINICAL TRIAL: NCT04734847
Title: Motor Cortical Neuromodulation in Women With Interstitial Cystitis/Bladder Pain Syndrome: Reducing Pain by Improving Brain and Muscle Activity
Brief Title: Motor Cortical Neuromodulation in Women With Interstitial Cystitis/Bladder Pain Syndrome
Acronym: IcBrainStim
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Jason Kutch, Associate Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APP-20-05139
Record Dates: First submitted 2021-01-27; First posted 2021-02-02 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Interstitial Cystitis; Bladder Pain Syndrome
Keywords: Chronic Pain; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Cystitis, Interstitial; Chronic Pain | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High-frequency rTMS (Active Comparator): Intensity: rTMS treatment intensity determined using resting motor threshold (RMT). Treatment will be delivered at 80% of the RMT.
  Site of Stimulation: Region of supplementary motor area (SMA) that regulates pelvic floor muscle activity. This target is defined in Montreal Neurological Institute (MNI) Coordinates of X=-2, Y=-16, and Z=68 mm.
  Frequency: 10 Hz.
  Duration: 20 Trains, 10 second duration, 50 second inter-train interval.
  Total number of pulses per session: 2000.
  Total number of session: 5 (one session per day for 5 consecutive days).
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)
- Sham rTMS (Sham Comparator): Identical to the High-frequency rTMS arm except delivered with an inert "sham" stimulation coil.
  Interventions: Device: Sham Repetitive Transcranial Magnetic Stimulation (Sham-rTMS)

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (rTMS) — Non-invasive magnetic stimulation of the brain
  Arms: High-frequency rTMS
Device: Sham Repetitive Transcranial Magnetic Stimulation (Sham-rTMS) — Device that appears identical to the active rTMS device, but does not produce any magnetic field and does not stimulate the brain.
  Arms: Sham rTMS

SUMMARY:
Interstitial Cystitis/Bladder Pain Syndrome (IC/BPS) is a common, chronic, and debilitating condition in women. Preliminary evidence suggests that IC/BPS pain can be reduced applying non-invasive repetitive transcranial magnetic stimulation (rTMS) to areas of the brain that regulate pelvic floor muscle activity. However, prior studies have examined rTMS in a very limited sample and have not examined changes in brain or pelvic floor muscle activity to determine the mechanism of rTMS for IC/BPS. This study is designed to directly address these limitations.

DETAILED DESCRIPTION:
Interstitial Cystitis/Bladder Pain Syndrome (IC/BPS) is a common, chronic, and debilitating condition in women. The underlying cause of IC/BPS remains unknown. We recently published the first functional magnetic resonance imaging (fMRI) study comparing brain function in women with IC/BPS to healthy women. We found that women with IC/BPS have altered resting activity in supplementary motor area (SMA). Specifically, these changes appear in a part of SMA that we have shown to control pelvic floor muscle activity. We call this part of SMA "pelvic-SMA". Our results provide the first potential explanation for extensive published reports of increased pelvic floor muscle activity in women with IC/BPS. We hypothesize that we are observing evidence of an important theory of chronic pain: motor cortical changes occur that are initially beneficial to increase protective muscle activity but are ultimately maladaptive and perpetuate pain. If this theory is true, it should be possible to reduce pain and muscle activity by improving brain activity. The proposed work is to do exactly that. Using non-invasive repetitive transcranial magnetic stimulation (rTMS) directed at pelvic-SMA, we aim to determine if we can reduce pain (Aim 1), improve resting brain activity (fMRI) and resting pelvic floor muscle electromyographic (EMG) activity in IC/BPS (Aim 2), and to link the pain reductions to fMRI/EMG improvements to develop a causal mediation model of IC/BPS symptoms (Aim 3). We will recruit 50 women with IC/BPS to participate in the study, and participants will be randomized to 2 groups of 25: high-frequency (active) or sham (inert). Our preliminary data suggest that high-frequency stimulation is the best stimulation protocol for reducing pain and improving pelvic-SMA activity and resting pelvic floor muscle activity. Our preliminary results agree with a large body of literature suggesting that high-frequency rTMS applied to motor cortex is the best stimulus paradigm to reduce pain, but our proposed work has the potential to greatly innovate the field of non-invasive brain stimulation for pain by providing a mechanism by which the stimulation can improve deficiencies in motor function in chronic pain patients.

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 18 years old.
2. Be female.
3. Have a diagnosis of IC/BPS by the referring physician, with urologic symptoms present a majority of the time during the most recent 3 months
4. Screen within standard limits for pelvic pain

Exclusion Criteria:

1. Symptomatic urethral stricture
2. On-going neurological conditions affecting the bladder or bowel
3. Active auto-immune or infectious disorders
4. History of cystitis caused by tuberculosis or radiation or chemotherapies
5. History of non-dermatologic cancer
6. Current major psychiatric disorders
7. Severe cardiac, pulmonary, renal, or hepatic disease
8. Conditions or the use of medical devices that are contraindications for either fMRI or rTMS procedures, including pregnancy, seizure disorders, or chronic headaches

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Longer-term Pain | Before first treatment to 3 weeks after last treatment
  Change in Visual Analog Scale of Pain. This scale ranges from 0 (no pain) to 10 (worst pain imaginable), so higher scores indicate more pain.
Shorter-term Pain | Before first treatment to 1 day later just before second treatment
  Change in Visual Analog Scale of Pain. This scale ranges from 0 (no pain) to 10 (worst pain imaginable), so higher scores indicate more pain.
Global Response Assessment | 3 weeks after last treatment
  Global Response Assessment (GRA)

SECONDARY OUTCOMES:
fALFF in Pelvic-SMA | One hour before and one hour after first treatment
  Change in fractional amplitude of low-frequency fluctuations (fALFF) derived from functional magnetic resonance imaging (fMRI) in targeted region of the brain (pelvic-SMA)
Pelvic floor muscle activity | Just before to between five and ten minutes after start of first treatment
  Change in activity of pelvic floor muscles as measured by electromyography (EMG). EMG is a physiological parameter measuring the electrical potential generated by a muscle, indicative of its activity. EMG is measured in micro-volts and then converted to percent change.

CONTACTS AND LOCATIONS:
Overall Officials: Jason J Kutch, PhD, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Johnson EV, Bachmann M, Yani MS, Eckel SP, Garcia GI, Rodriguez LV, Kutch JJ. Reducing pain by improving brain and muscle activity with motor cortical neuromodulation in women with interstitial cystitis/bladder pain syndrome: a study protocol for a randomized controlled trial. Trials. 2024 Sep 12;25(1):609. doi: 10.1186/s13063-024-08450-w. PMID 39261949